CLINICAL TRIAL: NCT03468270
Title: Pain Coping Strategies in Children With Cerebral Palsy
Brief Title: Pain Coping Strategies in Children With CP
Status: Completed | Type: Observational
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Other Study IDs: COPING
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Palsy; Pain
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe pain coping strategies and their evolution in children and adolescent with cerebral palsy.

DETAILED DESCRIPTION:
Towards the end of the 20th century, Lazarus and Folkmann developed the concept that the individual provides "cognitive and behavioral efforts to control, reduce or tolerate the internal or external demands that threaten or exceed his or her resources". These cognitive and behavioral efforts are grouped under the term "coping", which describes a process rather than personality traits or abilities. Coping is not about controlling stress but about diminishing, avoiding, tolerating or accepting it.

The pain, "unpleasant sensory and emotional experience related to a bodily injury", aims to warn the individual that the integrity of his body is threatened, and is thus a real "stressor". It will lead to the choice of coping strategies, which depends in part on the characteristics of the individual (his beliefs, stress endurance, anxiety propensity) and environmental variables (characteristics of the painful situation, social support and emotional connections, information about the threatening situation). Many studies have shown that the strategies used to cope with chronic pain in adults and children play a major role in the adjustment of patients to their pathology, in terms of emotional distress, disability, and quality of life. The different types of strategies have been widely studied in the literature in so-called "typical" children. Active strategies classically found in pediatrics are distraction, cognitive self-instruction, and problem solving. These active strategies are said to be positive because they have been proven to help children manage pain more effectively than passive strategies such as catastrophism, helplessness, or seeking social support, which are dysfunctional because they are not focused on the problem and increase the negative consequences associated with pain.

This study is about children with cerebral palsy (CP) because the great variability and complexity of the manifestations of the pathology and the therapeutic treatment make it that there is a big risk for the child to experience pain, with a prevalence of pain ranging from 60% to 73%, depending on the evaluation methods. Research has done a great deal in recent years to improve the assessment and management of inborn or induced pain in children with disabilities, with many validated recommendations, even though this still appears to be a neglected comorbidity in PC. However, coping strategies of PC children with pain have never been studied. The purpose of this work is to describe these strategies in PC children and adolescents, as well as their evolution.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnostic of cerebral palsy
* GMFCS I, II, III, IV
* Oral language skills with syntactic abilities

Exclusion Criteria:

* Acute pain episode
* severe cognitive impairment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients were recruited in the services of 2 French Red Cross Physical Medicine and Rehabilitation Centers in France. All parents and children were informed orally about the procedure, and parental consent as the child's consent was obtained in writing.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
PPCI-F (Pediatric Pain and Coping inventory - French) | At inclusion
  Coping strategies used to face pain are measured by the French version of the PPCI. This scale leads to 4 subscores, corresponding to 4 different strategies.

SECONDARY OUTCOMES:
SPQ (Structured Pain Questionnaire) | At inclusion
  This questionnaire assesses the location and frequency of pain episodes (<1 time / month, 1 time / month, 2-3 times / month, 1 time / week, 2-6 times / week, each day), their duration (<4 weeks, 4 weeks, 3 months,> 3 months) and pain intensity (0 to 100 on scoring scale).
Evolution of PPCI-F scores according to age. | At inclusion
  The evolution of the coping strategies used according to the age of the patient is assessed by the Spearman correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix rouge française Centre Médico-Chirurgical de Réadaptation des Massues, Lyon, France

IPD SHARING:
Plan to Share IPD: No